CLINICAL TRIAL: NCT01830816
Title: Phase 1/1b Pharmacokinetics Study of Oral MLN9708 in Patients With Relapsed/Refractory Multiple Myeloma and Advanced Solid Tumors With Normal Renal Function or Severe Renal Impairment
Brief Title: Pharmacokinetics Study of Oral Ixazomib (MLN9708) in Relapsed/Refractory Multiple Myeloma and Advanced Solid Tumors Participants With Normal Renal Function or Severe Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C16015; U1111-1158-2763 (Registry Identifier: WHO); 165055 (Registry Identifier: HC-CTD)
Record Dates: First submitted 2013-04-04; First posted 2013-04-12 (Estimated); Results first posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-03

CONDITIONS: Multiple Myeloma; Advanced Solid Tumors
Keywords: Drug Therapy
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Normal Renal Function: Ixazomib (Experimental): In the 15 day period that constitutes Part A of the trial, participants received a single oral dose of ixazomib 3.0 mg capsules. Participants from Part A had the option of continuing the study by participating in Part B, where they received ixazomib (4, 3, or 2.3 mg per protocol) capsules, orally on Days 1, 8, and 15 of each 28-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Ixazomib
- Severe Renal Impairment: Ixazomib (Experimental): In the 15 day period that constitutes Part A of the trial, participants received a single oral dose of ixazomib 3.0 mg capsules. Participants from Part A had the option of continuing the study by participating in Part B, where they received ixazomib (4, 3, or 2.3 mg per protocol) capsules, orally on Days 1, 8, and 15 of each 28-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Ixazomib
- End-stage Renal Disease: Ixazomib (Experimental): In the 15 day period that constitutes Part A of the trial, participants received a single oral dose of ixazomib 3.0 mg capsules. Participants from Part A had the option of continuing the study by participating in Part B, where they received ixazomib (4, 3, or 2.3 mg per protocol) capsules, orally on Days 1, 8, and 15 of each 28-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Ixazomib

INTERVENTIONS:
Drug: Ixazomib — Ixazomib capsules
  Other Names: MLN9708

SUMMARY:
The purpose of this study is to characterize the single-dose pharmacokinetic (PK) parameters of ixazomib (MLN9708) in cancer participants with either normal renal function or severe renal impairment (RI), including participants with end-stage renal disease (ESRD).

DETAILED DESCRIPTION:
The drug tested in this study was called ixazomib (MLN9708). Ixazomib was administered to participants with cancer and either normal renal function or severe renal impairment, including end-stage renal disease (ESRD) requiring hemodialysis. This study characterized the PK, safety and efficacy of ixazomib.

The study enrolled 41 participants (37 multiple myeloma and 4 advanced solid tumor). The study was conducted in 2 parts, Part A and Part B. Participants were enrolled to receive:

* Ixazomib 3.0 mg

In Part A, all participants were asked to take one 3 mg ixazomib capsule, orally on Day 1. Participants who tolerated ixazomib in Part A had the option of continuing the study by participating in Part B. In Part B, participants received ixazomib (4, 3, or 2.3 mg per protocol) on Days 1, 8, and 15 of each 28-day cycle until participants experienced disease progression or unacceptable toxicity.

This multicenter trial was conducted at 6 study sites in the United States and Canada. The overall time to participate in this study was 435 days. Participants made multiple scheduled visits to the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants 18 years or older
* Participants with multiple myeloma (MM) diagnosed according to standard criteria or participants with a diagnosis of an advanced malignant solid tumor for which standard, curative, or life prolonging treatment does not exist or is no longer effective. Participants with multiple myeloma must have had at least 1 prior therapy
* A calculated creatinine clearance (CrCl) that meets entry criteria for enrollment (i.e., calculated CrCl either ≥ 90 mL/min for normal renal function or < 30 mL/min for severe renal impairment)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Female participants who are post menopausal, surgically sterile, or agree to practice 2 effective methods of contraception through 90 days after the last dose of study drug or agree to practice true abstinence
* Male participants who agree to practice effective barrier contraception through 90 after the last dose of study drug or agree to practice true abstinence
* Voluntary written informed consent
* Suitable venous access

Exclusion Criteria:

* Female participants who are pregnant or lactating and breastfeeding
* Failure to have recovered from clinically significant effects of prior chemotherapy (defined as toxicity greater than Grade 1 with the exception of alopecia)
* Major surgery or radiotherapy within 14 days before study drug administration
* Dexamethasone (or equivalent systemic steroid) higher than physiologic dosing within 7 days before study drug administration
* Central nervous system involvement
* Infection requiring IV antibiotic therapy or other serious infection within 14 days prior to first dose of study drug
* Diagnosis of Waldenstrom's macroglobulinemia, POEMS (polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes) syndrome, plasma cell leukemia, myeloproliferative syndrome, or primary amyloidosis (with the exception of patients in whom amyloidosis has been documented as a complication of MM, who will be evaluated on a case-by-case basis for trial participation)
* Systemic treatment with strong and moderate inhibitors of Cytochrome P1A2 (CYP1A2), strong and moderate inhibitors of Cytochrome P3A (CYP3A), or clinically significant CYP3A inducers or use of Ginkgo biloba or St. John's wort within 14 days before the first dose of study drug
* Evidence of uncontrolled cardiovascular conditions
* Ongoing or active infection, or known human immunodeficiency virus (HIV) positive
* Comorbid systemic illness or psychiatric illness that could interfere with study completion
* Known allergy to study medications
* Inability to swallow oral medication or condition that could interfere with oral absorption or tolerance of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-09-16 (Actual); Primary Completion 2015-03-03 (Actual); Study Completion 2016-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (11):
- United States (10):
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Illinois Cancer Care, Peoria, Illinois
  - University of Kansas Cancer Center, Clinical Research Center, Fairway, Kansas
  - University of Maryland, Baltimore, Maryland
  - Mount Sinai Medical Center, New York, New York
  - University of Oklahoma Peggy and Charles Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - Mary Crowley Cancer Research Centers Medical City, Dallas, Texas
  - Institute of Oncology Hematology Biomedical Research, Laredo, Texas
  - University of Texas Health Science Center San Antonio, San Antonio, Texas
- University Health Network, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 6 investigative sites in the United States and Canada from 16 September 2013 up to 18 November 2016.
Pre-assignment Details: Participants with a diagnosis of relapsed or refractory multiple myeloma (RRMM) or advanced solid tumors who had normal renal function or severe renal impairment including end-stage renal disease requiring hemodialysis (ESRD) were enrolled to receive ixazomib orally in the study.
Groups:
- Normal Renal Function: Ixazomib; Severe Renal Impairment: Ixazomib; End-stage Renal Disease: Ixazomib: Ixazomib 3.0 mg, capsule, orally on Day 1 of Part A (15-day PK cycle) and on Days 1, 8, and 15 of each 28-day cycle in Part B (4.0, 3.0, or 2.3 mg per protocol) until disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Normal Renal Function: Ixazomib | Severe Renal Impairment: Ixazomib | End-stage Renal Disease: Ixazomib
Started | 20 | 14 | 7
Pharmacokinetic-Evaluable Population | 18 (Participants are considered to have completed study treatment if they are PK evaluable.) | 14 | 6
Completed | 0 | 0 | 0
Not Completed | 20 | 14 | 7
Not completed — Progressive Disease | 12 | 7 | 7
Not completed — Adverse Event | 3 | 4 | 0
Not completed — Study Terminated by Sponsor | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Symptomatic Deterioration | 1 | 0 | 0
Not completed — Reason not Specified | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population is defined as participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Renal Function: Ixazomib | Severe Renal Impairment: Ixazomib | End-stage Renal Disease: Ixazomib | Total
Number analyzed (Participants) | 20 | 14 | 7 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (9.01) | 72.1 (7.35) | 61.3 (12.65) | 61.7 (12.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 3 | 25
  Male | 10 | 2 | 4 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 4
  Not Hispanic or Latino | 19 | 10 | 6 | 35
  Not Reported | 0 | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 13 | 11 | 3 | 27
  Black or African American | 6 | 3 | 3 | 12
  Asian | 0 | 0 | 1 | 1
  Not Reported | 1 | 0 | 0 | 1
Height [Mean (Standard Deviation); unit: cm] — Population: Number analyzed is the number of participants with data available for height.
  cm
    number analyzed (Participants) | 20 | 14 | 5 | 39
    (all) | 173.2 (11.28) | 160.8 (8.49) | 160.3 (9.61) | 167.1 (11.76)
Weight [Mean (Standard Deviation); unit: kg] | 98.1 (27.66) | 60.7 (14.70) | 86.0 (27.11) | 83.3 (28.85)

OUTCOME MEASURES:

1. Primary Outcome: Unbound Cmax: Unbound Maximum Observed Plasma Concentration for Ixazomib
Time Frame: Part A, Day 1: Predose and at multiple timepoints (up to 336 hours) post-dose
Population: Pharmacokinetic (PK) evaluable population was defined as participants who received protocol-specified single dose in Part A; did not receive any excluded concomitant medications through the completion of PK sampling; and had sufficient concentration-time data to permit reliable estimation of PK parameters by non-compartmental analysis methods.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Normal Renal Function: Ixazomib | Severe Renal Impairment: Ixazomib | End-stage Renal Disease: Ixazomib
Number analyzed (Participants) | 18 | 14 | 6
ng/mL | 0.300 (0.247944) | 0.478 (0.599519) | 0.213 (0.136696)

2. Primary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Ixazomib
Time Frame: Part A, Day 1: Predose and at multiple timepoints (up to 336 hours) post-dose
Population: PK evaluable population was defined as participants who received protocol-specified single dose in Part A; did not receive any excluded concomitant medications through the completion of PK sampling; and had sufficient concentration-time data to permit reliable estimation of PK parameters by non-compartmental analysis methods.
Measure: Median (Full Range); unit: hours
Arm/Group | Normal Renal Function: Ixazomib | Severe Renal Impairment: Ixazomib | End-stage Renal Disease: Ixazomib
Number analyzed (Participants) | 18 | 14 | 6
hours | 1.0400 [0.467 to 4.000] | 1.0000 [0.450 to 1.500] | 1.2500 [0.983 to 7.000]

3. Primary Outcome: Unbound AUClast: Unbound Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Ixazomib
Time Frame: Part A, Day 1: Predose and at multiple timepoints (up to 336 hours) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Normal Renal Function: Ixazomib | Severe Renal Impairment: Ixazomib | End-stage Renal Disease: Ixazomib
Number analyzed (Participants) | 15 | 10 | 6
hr*ng/mL | 6.637 (4.8022) | 9.249 (6.2618) | 8.925 (5.7995)

4. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse Event is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: From signing of first dose of study drug up to the 30 days after the last dose of study drug (approximately up to 885 days)
Population: Safety population is defined as participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Normal Renal Function: Ixazomib | Severe Renal Impairment: Ixazomib | End-stage Renal Disease: Ixazomib
Number analyzed (Participants) | 20 | 14 | 7
participants | 19 | 14 | 6

5. Secondary Outcome: Percentage of Participants With Overall Response (OR) in Relapsed/Refractory Multiple Myeloma (RRMM) Participants
Description: Overall response rate defined as percentage of relapsed/refractory multiple myeloma participants who achieved partial response (PR), complete response (CR) and very good partial response (VGPR) according to International Myeloma Working Group Criteria. PR=>50% reduction of serum M-protein and reduction in 24 hours urinary M-protein by >90% or <200 mg/24 h. If serum and urine M-protein are unmeasurable, >50% decrease in difference between involved and uninvolved free light chain levels in place of M-protein criteria. If serum and urine M-protein and serum free light assay are not measurable, >50% reduction in plasma cells in place of M-protein, provided baseline bone marrow plasma cell >0%; CR=negative immunofixation on serum and urine and disappearance of any soft tissue plasmacytomas and <5% plasma cells in bone marrow; VGPR=serum and urine M-protein detectable by immunofixation but not on electrophoresis or > 90% reduction in serum M-protein plus urine M-protein level <100 mg/24 h.
Time Frame: Day 1 of every other cycle from cycle 1 (each cycle of 28 days) up to progression of disease (approximately up to 855 days)
Population: Response evaluable is defined as participants who received at least 1 cycle of ixazomib treatment in Part B and at least 1 post-baseline response assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Normal Renal Function: Ixazomib; Severe Renal Impairment: Ixazomib; End-stage Renal Disease: Ixazomib: After part A the participant has the option to participate in Part B start with ixazomib capsules, orally on Days 1, 8, and 15 of each 28-day cycle until disease progression or unacceptable toxicity.
Arm/Group | Normal Renal Function: Ixazomib | Severe Renal Impairment: Ixazomib | End-stage Renal Disease: Ixazomib
Number analyzed (Participants) | 14 | 11 | 4
percentage of participants | 29 [8 to 58] | 18 [2 to 52] | 0 [NA to NA] — No participant had overall response.

6. Secondary Outcome: Duration of Response (DOR) in RRMM Participants
Description: DOR was defined as time from date of first documentation of a PR or better to date of first documentation of progressive disease (PD) for responders. Increase of >25% from lowest response value in any one or more of following: Serum M-component and/or (absolute increase must be >0.5 g/dL); Urine M-component and/or (the absolute increase must be >200 mg/24 h); difference between involved and uninvolved free light chain (FLC) levels and the absolute increase must be > 10 mg/dL; Bone marrow plasma cell percentage; absolute percentage must be > 5%; Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in size of existing bone lesions or soft tissue plasmacytomas; Development of hypercalcaemia (corrected serum calcium > 11.5 mg/dL or 2.65 mmol/L) that can be attributed solely to the plasma cell proliferative disorder. Responders without PD were censored at the date of the last response assessment that was stable disease (SD) or better.
Time Frame: as for outcome 5
Population: Response evaluable population is defined as participants who received at least 1 cycle of Ixazomib treatment in Part B and at least 1 post-baseline response assessment. Here, number of participants analyzed is the participants who had confirmed response.
Measure: Median (Full Range); unit: days
Arm/Group | Normal Renal Function: Ixazomib | Severe Renal Impairment: Ixazomib | End-stage Renal Disease: Ixazomib
Number analyzed (Participants) | 4 | 2 | 0
days | 134 [72 to 233] | 225 [225 to 225] |

ADVERSE EVENTS:
Time Frame: From signing of first dose of study drug up to the 30 days after the last dose of study drug (approximately up to 885 days)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Groups:
- Normal Renal Function: Ixazomib: Ixazomib 3.0 mg, capsules, orally once on Day 1 of part A of 15 days followed by ixazomib 4 mg, capsules, orally on Days 1, 8, and 15 of each 28-day cycle in normal renal function participants until disease progression or unacceptable toxicity in part B.
  Dose modification of 3 or 2.3 mg was administered per protocol dose modification guidelines.
- Severe Renal Impairment: Ixazomib: Ixazomib 3.0 mg, capsules, orally once on Day 1 of part A of 15 days followed by ixazomib 4 mg, capsules, orally on Days 1, 8, and 15 of each 28-day cycle in severe renal impairment participants until disease progression or unacceptable toxicity in part B.
  Dose modification of 3 or 2.3 mg was administered per protocol dose modification guidelines.
- End-stage Renal Disease: Ixazomib: Ixazomib 3.0 mg, capsules, orally once on Day 1 of part A of 15 days followed by ixazomib 4 mg, capsules, orally on Days 1, 8, and 15 of each 28-day cycle in end-stage renal disease participants until disease progression or unacceptable toxicity in part B.
  Dose modification of 3 or 2.3 mg was administered per protocol dose modification guidelines.
Arm/Group | Normal Renal Function: Ixazomib | Severe Renal Impairment: Ixazomib | End-stage Renal Disease: Ixazomib
Serious Adverse Events (participants affected / at risk) | 3/20 | 6/14 | 3/7
Other Adverse Events (participants affected / at risk) | 19/20 | 14/14 | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Normal Renal Function: Ixazomib (N=20) | Severe Renal Impairment: Ixazomib (N=14) | End-stage Renal Disease: Ixazomib (N=7)
Bronchitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 — One treatment-emergent death occurred during treatment with ixazomib in severe renal impairment arm group and is not related.
Bacteraemia (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Skin infection (Infections and infestations) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 — One treatment-emergent death occurred during treatment with ixazomib in end stage renal disease arm group and is not related.
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 — One treatment-emergent death occurred during treatment with ixazomib in severe renal impairment arm group and is related.
Gastrooesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal Renal Function: Ixazomib (N=20) | Severe Renal Impairment: Ixazomib (N=14) | End-stage Renal Disease: Ixazomib (N=7)
Diarrhoea (Gastrointestinal disorders) | 8 | 6 | 1
Nausea (Gastrointestinal disorders) | 7 | 5 | 2
Vomiting (Gastrointestinal disorders) | 6 | 5 | 2
Constipation (Gastrointestinal disorders) | 6 | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 5 | 6 | 1
Oedema peripheral (General disorders) | 2 | 4 | 0
Pyrexia (General disorders) | 2 | 2 | 0
Chest discomfort (General disorders) | 2 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 (1) | 4 (4) | 1 (1)
Headache (Nervous system disorders) | 4 (6) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (4) | 2 (3) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 2 (3) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (4) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Weight increased (Investigations) | 3 | 3 | 0
Platelet count decreased (Investigations) | 1 | 3 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 1 | 0
Weight decreased (Investigations) | 0 | 2 | 0
Ammonia increased (Investigations) | 0 | 0 | 1
Creatinine renal clearance increased (Investigations) | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 5 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 3 | 0
Fungal skin infection (Infections and infestations) | 2 | 0 | 0
Herpes virus infection (Infections and infestations) | 1 | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (3) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Mood altered (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Cataract (Eye disorders) | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 1 | 0
Middle ear effusion (Ear and labyrinth disorders) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0
Cardiac disorders (Cardiac disorders) | 2 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.